CLINICAL TRIAL: NCT05081024
Title: Establishing a ctDNA Biomarker to Improve Organ Preserving Strategies in Patients With Rectal Cancer
Status: Recruiting | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Natera, Inc. (Industry)
Responsible Party: Principal Investigator, Adel Kardosh M.D., Ph.D., Principal Investigator, OHSU Knight Cancer Institute
Other Study IDs: STUDY00022247; NCI-2021-08733 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00022247 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2021-09-07; First posted 2021-10-18 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Rectal Adenocarcinoma; Stage II Rectal Cancer AJCC v8; Stage IIA Rectal Cancer AJCC v8; Stage IIB Rectal Cancer AJCC v8; Stage IIC Rectal Cancer AJCC v8; Stage III Rectal Cancer AJCC v8; Stage IIIA Rectal Cancer AJCC v8; Stage IIIB Rectal Cancer AJCC v8; Stage IIIC Rectal Cancer AJCC v8
MeSH Terms: conditions — Rectal Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (biospecimen collection, medical record review): Patients undergo collection of blood samples at baseline (before any neoadjuvant therapy), every 2 months while undergoing TNT, and then every 3 months for up to 3 years after completion of TNT. Patients' medical records are also reviewed. Patients may undergo collection of tissue sample if an archival tissue sample is not available.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Other: Electronic Health Record Review

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood and/or tissue samples
  Other Names: Biological Sample Collection
Other: Electronic Health Record Review — Medical records are reviewed

SUMMARY:
This study measures the levels of circulating tumor DNA (ctDNA) in patients with stage II-III rectal cancer before, during, and after treatment to find out if the presence or absence of ctDNA in patient's blood using the Signatera test can be used to gauge how different treatments may affect rectal cancer. ctDNA is DNA from the rectal cancer that is circulating in the blood. The purpose of this study is to understand if the way rectal tumors respond to standard treatment can be associated with varying levels of ctDNA.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the percentage of participants that achieve complete clinical response.

SECONDARY OBJECTIVES:

I. To assess circulating tumor deoxyribonucleic acid (ctDNA) status among participants receiving total neoadjuvant therapy (TNT).

II. To assess molecular residual disease (MRD i.e., ctDNA status). III. To assess the rate of transabdominal surgery. IV. To assess the rate pathological complete response after surgery. V. To assess the rate of watch and -wait (W&W) after TNT. VI. To assess disease-free survival (DFS). VII. To assess overall survival (OS).

EXPLORATORY OBJECTIVES:

I. To characterize ctDNA clearance or non-clearance patterns during TNT. II. To correlate ctDNA levels with a participant's pathological features. III. To preliminary assess the prognostic performance of ctDNA levels in relation to participant's clinical outcome.

OUTLINE:

Patients undergo collection of blood samples at baseline (before any neoadjuvant therapy), every 2 months while undergoing TNT, and then every 3 months for up to 3 years after completion of TNT. Patients' medical records are also reviewed. Patients may undergo collection of tissue sample if an archival tissue sample is not available.

ELIGIBILITY:
Inclusion Criteria:

* Participant must provide written informed consent before any study-specific procedures or interventions are performed
* Participants aged >= 18 years
* Pathologically-confirmed stage II or III primary adenocarcinoma of the rectum:

  * T3N0M0 - T4bN2M0

Exclusion Criteria:

* Has radiologic evidence of distant metastases at the time of screening/enrollment
* Has received prior treatment for their rectal adenocarcinoma
* Requires or has received blood transfusion within 1 month of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage II-III rectal adenocarcinoma at Oregon Health & Science University (OHSU), its affiliated community oncology (CHO) site, or collaborating research site
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2026-09-03 (Estimated); Study Completion 2026-09-03 (Estimated)

PRIMARY OUTCOMES:
Complete clinical response (cCR) | From time of treatment start up to date of completing total neoadjuvant therapy (TNT), up to 3 months.
  cCR following TNT will be analyzed using the TNT analysis set. Proportions of participants that achieved cCR will be calculated and the exact 95% confidence interval (CI) will be presented.

SECONDARY OUTCOMES:
Positive circulating tumor deoxyribonucleic acid (ctDNA) | From date of baseline measure of ctDNA (i.e., number of mutant molecules per mL) to date of until the date of first documented progression, up to 3 years.
  The proportion of ctDNA positive participants (at baseline, throughout TNT, and follow-up) and its exact 95% CI will be evaluated using the ctDNA analysis set. Where appropriate, sub-analyses will be conducted using populations that underwent surgery or were monitored using a watch and wait (W&W) strategy.
Positive ctDNA after completing TNT | From date of baseline measure of ctDNA (i.e., number of mutant molecules per mL) to date of until the date of first documented progression, up to 3 years
  The proportion of ctDNA positive participants (at baseline, throughout TNT, and follow-up) and its exact 95% CI will be evaluated using the ctDNA analysis set. Where appropriate, sub-analyses will be conducted using populations that underwent surgery or were monitored using a W&W strategy.
Rate of transabdominal surgery | Up to 3 years following completion of TNT
  Will be evaluated using the TNT analysis set. The corresponding exact 95% CI will also be presented.
Rate of pathological complete response (pCR) | From start of treatment until completion of surgery, up to 3 years.
  Will be evaluated using the TNT analysis set. The corresponding exact 95% CI will also be presented.
Rate of watch and wait strategy | Up to 3 years following completion of TNT
  Will be evaluated using the TNT analysis set. The corresponding exact 95% CI will also be presented.
Disease-free survival | Time between the date of surgery (or W&W population, the date of completing TNT) and the date of local or metastatic recurrence or death from any cause, assessed up to 3 years following completion of TNT
  Will be estimated using the Kaplan-Meier method.
Overall survival | Time between the date of signed consent to the date of death from any cause, assessed up to 3 years following completion of TNT
  Will be estimated using the Kaplan-Meier method.

OTHER OUTCOMES:
ctDNA status | From date of baseline measure of ctDNA (i.e., number of mutant molecules per mL) to date of until the date of first documented progression, up to 3 years
  positive versus negative results per test results
Positive ctDNA by clinical characteristics | From date of baseline measure of ctDNA to date of recurrence or death from any cause, assessed up to 3 years following completion of TNT
  association or recurrence on ctDNA test and standard imaging
Sensitivity | From date of baseline measure of ctDNA to date of recurrence or death from any cause, assessed up to 3 years following completion of TNT
  Sensitivity and specificity will be calculated using complete clinical response (yes versus [vs.] no), or tumor recurrence (yes vs. no) as reference standard.
Specificity | From date of baseline measure of ctDNA to date of recurrence or death from any cause, assessed up to 3 years following completion of TNT
  Sensitivity and specificity will be calculated using complete clinical response (yes vs. no), or tumor recurrence (yes vs. no) as reference standard.

CONTACTS AND LOCATIONS:
Overall Officials: Adel Kardosh, M.D.,Ph.D., Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Fred Hutch, Seattle, Washington